CLINICAL TRIAL: NCT01091103
Title: A Study Of Continuous Oral Dosing Of A Novel Antiandrogen Mdv3100, In Castration-resistant Bone Metastatic Prostate Cancer Patients Evaluating The Tumor Micro-enviroment
Brief Title: Determine Effect of Enzalutamide (MDV3100) on the Androgen Signaling Pathway in Correlation With the Anti-tumor Effects of Enzalutamide
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Pfizer (Industry)
Collaborators: Astellas Pharma Inc (Industry); Medivation LLC, a wholly owned subsidiary of Pfizer Inc. (Industry)
Responsible Party: Sponsor
Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CRPC-MDA-1; C3431017 (Other: Alias Study Number)
Record Dates: First submitted 2010-03-19; First posted 2010-03-23 (Estimated); Results first posted 2014-11-17 (Estimated); Last update posted 2018-10-23 (Actual); Status verified 2018-10

CONDITIONS: Metastatic Progressive Castration-resistant Prostate Cancer
MeSH Terms: interventions — enzalutamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Enzalutamide (Experimental): Participants received enzalutamide 160 mg, administered as four 40-mg capsules, once per day by mouth. Study drug treatment continued until disease progression, unacceptable toxicity, or withdrawal.
  Interventions: Drug: Enzalutamide

INTERVENTIONS:
Drug: Enzalutamide
  Other Names: MDV3100

SUMMARY:
This study is being conducted to determine the effect of enzalutamide on the androgen signaling pathway in correlation with the anti-tumor effects of enzalutamide to identify potential predictors of response or resistance to therapy.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed prostate cancer
* Presence of metastatic disease to the bone
* Ongoing androgen deprivation therapy

Exclusion Criteria:

* Severe concurrent disease
* Metastases in the brain

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 60 (Actual)
Dates: Start 2010-02-18 (Actual); Primary Completion 2012-02-29 (Actual); Study Completion 2013-08-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer; Medical Monitor, Study Director — Medivation, Inc.
Locations (1):
- MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- [Derived] Efstathiou E, Titus M, Wen S, Hoang A, Karlou M, Ashe R, Tu SM, Aparicio A, Troncoso P, Mohler J, Logothetis CJ. Molecular characterization of enzalutamide-treated bone metastatic castration-resistant prostate cancer. Eur Urol. 2015 Jan;67(1):53-60. doi: 10.1016/j.eururo.2014.05.005. Epub 2014 May 29. PMID 24882673

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Single center clinical trial
Groups:
- Enzalutamide: Participants received enzalutamide 160 mg, administered as four 40-mg capsules, once per day by mouth.
Period: Overall Study
Arm/Group | Enzalutamide
Started | 60
Completed | 56 (Patients on study drug and completed Week 9 visit assessments.)
Not Completed | 4
Not completed — Adverse Event | 1
Not completed — Progressive Disease | 3

BASELINE CHARACTERISTICS:
Arm/Group | Enzalutamide
Number analyzed (Participants) | 60
Age, Continuous [Mean (Standard Deviation); unit: years] | 67.9 (9.99)
Age, Customized [Number; unit: years]
  < 55 | 6
  55 to < 65 | 17
  65 to < 75 | 18
  >= 75 | 19
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 60

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Bone Marrow Testosterone
Description: Bone marrow biopsies were performed at the Day 1 visit prior to initiation of enzalutamide administration. Repeat bone marrow biopsies were performed at the Week 9 visit. If a repeat bone marrow was not performed at the Week 9 visit or if a patient discontinued the study before the Week 9 visit, a bone marrow biopsy was obtained at the Safety Follow-up visit.
  Assessment of intratumoral testosterone was assessed by liquid chromatography mass spectrometry.
Time Frame: Baseline, Week 9
Population: Participants who received any amount of enzalutamide and had bone marrow testosterone measurements at baseline and at least 1 post-baseline assessment. Note that the documentation of bone marrow involvement with cancer was not required.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Enzalutamide
Number analyzed (Participants) | 31
ng/mL | 0.05 (0.072)

2. Secondary Outcome: Percentage of Participants at Week 9 With a Response in Prostate-Specific Antigen (PSA)
Description: Serum samples for measurement of PSA levels were obtained at baseline prior to initiation of enzalutamide administration and at the Week 9 visit.
Time Frame: Baseline, Week 9
Population: Participants who received any amount of enzalutamide and had PSA values at baseline and at the Week 9 Visit.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Enzalutamide
Number analyzed (Participants) | 56
percentage of participants
  >=50% Reduction in PSA from Baseline | 41.1 [28.1 to 55.0]
  >=90% Reduction in PSA from Baseline | 21.4 [11.6 to 34.4]

3. Primary Outcome: Change From Baseline in Bone Marrow Dihydrotestosterone
Description: Bone marrow biopsies were performed at the Day 1 visit prior to initiation of enzalutamide administration. Repeat bone marrow biopsies were performed at the Week 9 visit. If a repeat bone marrow was not performed at the Week 9 visit or if a patient discontinued the study before the Week 9 visit, a bone marrow biopsy was obtained at the Safety Follow-up visit.
  Assessment of intratumoral dihydrotestosterone was assessed by liquid chromatography mass spectrometry.
Time Frame: Baseline, Week 9
Population: Participants who received any amount of enzalutamide and had bone marrow dihydrotestosterone measurements at baseline and at least 1 post-baseline assessment. Note that the documentation of bone marrow involvement with cancer was not required.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Enzalutamide
Number analyzed (Participants) | 31
ng/mL | 0.00 (0.022)

4. Primary Outcome: Change From Baseline in Bone Marrow Testosterone at Week 9 by Prostate-Specific Antigen (PSA) Response Status
Description: Bone marrow biopsies were performed at the Day 1 visit prior to initiation of enzalutamide administration. Repeat bone marrow biopsies were performed at the Week 9 visit. If a repeat bone marrow was not performed at the Week 9 visit or if a patient discontinued the study before the Week 9 visit, a bone marrow biopsy was obtained at the Safety Follow-up visit. Assessment of intratumoral testosterone was assessed by liquid chromatography mass spectrometry.
  Serum samples for measurement of PSA levels were obtained at baseline prior to initiation of enzalutamide administration and at the Week 9 visit.
  The change from baseline in bone marrow testosterone levels at Week 9 was correlated with PSA response status at Week 9.
Time Frame: Baseline, Week 9
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: ng/mL
Groups:
- Enzalutamide, PSA Responders at Week 9: PSA responders are defined by a greater than or equal to 50% reduction from baseline in PSA at Week 9
- Enzalutamide, PSA Non-Responders at Week 9: PSA non-responders are defined by a less than 50% reduction from baseline in PSA at Week 9
Arm/Group | Enzalutamide, PSA Responders at Week 9 | Enzalutamide, PSA Non-Responders at Week 9
Number analyzed (Participants) | 13 | 18
ng/mL | 0.05 (0.107) | 0.05 (0.034)
Statistical Analysis 1: Comparison: Enzalutamide, PSA Responders at Week 9 vs Enzalutamide, PSA Non-Responders at Week 9; Test type: Superiority or Other; p = 0.9427, t-test, 2 sided — The p-value was not adjusted for multiplicity

5. Primary Outcome: Change From Baseline in Bone Marrow Dihydrotestosterone at Week 9 by Prostate-Specific Antigen (PSA) Response Status
Description: Bone marrow biopsies were performed at the Day 1 visit prior to initiation of enzalutamide administration. Repeat bone marrow biopsies were performed at the Week 9 visit. If a repeat bone marrow was not performed at the Week 9 visit or if a patient discontinued the study before the Week 9 visit, a bone marrow biopsy was obtained at the Safety Follow-up visit. Assessment of intratumoral dihydrotestosterone was assessed by liquid chromatography mass spectrometry.
  Serum samples for measurement of PSA levels were obtained at baseline prior to initiation of enzalutamide administration and at the Week 9 visit.
  The change from baseline in bone marrow dihydrotestosterone levels at Week 9 was correlated with PSA response status at Week 9.
Time Frame: Baseline, Week 9
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Enzalutamide, PSA Responders at Week 9 | Enzalutamide, PSA Non-Responders at Week 9
Number analyzed (Participants) | 13 | 18
ng/mL | -0.01 (0.034) | 0.00 (0.000)
Statistical Analysis 1: Comparison: Enzalutamide, PSA Responders at Week 9 vs Enzalutamide, PSA Non-Responders at Week 9; Test type: Superiority or Other; p = 0.3370, t-test, 2 sided — The p-value was not adjusted for multiplicity

6. Secondary Outcome: Median Time to Study Drug Discontinuation
Description: Exposure to study drug through the data cutoff of 26AUG2011 only. Fifteen participants (25.0%) were still on study drug as of the data cut-off date and were censored at this date.
Time Frame: Duration of study treatment through the data cutoff, up to 3 years.
Population: All participants who received any amount of enzalutamide. Fifteen (25.0%) participants were still on study drug as of the data cutoff date and were censored at the data cutoff date.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Enzalutamide
Number analyzed (Participants) | 60
months | 5.0 [3.6 to 6.0]

7. Secondary Outcome: Change From Baseline in Urinary N-Telopeptide
Description: Samples for measurement of urinary N-telopeptide were collected at baseline prior to initiation of enzalutamide administration and at Week 5.
Time Frame: Baseline, Week 5
Population: Participants who received any amount of enzalutamide and had urinary N-telopeptide measurements at baseline and at Week 5.
Measure: Mean (Standard Deviation); unit: mmol/mmol creatinine
Arm/Group | Enzalutamide
Number analyzed (Participants) | 59
mmol/mmol creatinine | 34.81 (137.361)

8. Secondary Outcome: Change From Baseline in Urinary N-Telopeptide
Description: Samples for measurement of urinary N-telopeptide were collected at baseline prior to initiation of enzalutamide administration and at Week 9.
Time Frame: Baseline, Week 9
Population: Participants who received any amount of enzalutamide and had urinary N-telopeptide measurements at baseline and at Week 9.
Measure: Mean (Standard Deviation); unit: mmol/mmol creatinine
Arm/Group | Enzalutamide
Number analyzed (Participants) | 55
mmol/mmol creatinine | 205.84 (1334.820)

9. Secondary Outcome: Change From Baseline in Urinary N-Telopeptide
Description: Samples for measurement of urinary N-telopeptide were collected at baseline prior to initiation of enzalutamide administration and at Week 17.
Time Frame: Baseline, Week 17
Population: Participants who received any amount of enzalutamide and had urinary N-telopeptide measurements at baseline and at Week 17.
Measure: Mean (Standard Deviation); unit: mmol/mmol creatinine
Arm/Group | Enzalutamide
Number analyzed (Participants) | 39
mmol/mmol creatinine | -0.92 (205.941)

10. Secondary Outcome: Change From Baseline in Urinary N-Telopeptide
Description: Samples for measurement of urinary N-telopeptide were collected at baseline prior to initiation of enzalutamide administration and at Week 25.
Time Frame: Baseline, Week 25
Population: Participants who received any amount of enzalutamide and had urinary N-telopeptide measurements at baseline and at Week 25.
Measure: Mean (Standard Deviation); unit: mmol/mmol creatinine
Arm/Group | Enzalutamide
Number analyzed (Participants) | 27
mmol/mmol creatinine | -18.96 (278.112)

11. Secondary Outcome: Change From Baseline in Urinary N-Telopeptide
Time Frame: Baseline, Week 33
Population: Participants who received any amount of enzalutamide and had urinary N-telopeptide measurements at baseline and at Week 33.
Measure: Mean (Standard Deviation); unit: mmol/mmol creatinine
Arm/Group | Enzalutamide
Number analyzed (Participants) | 14
mmol/mmol creatinine | -89.36 (363.140)

12. Secondary Outcome: Change From Baseline in Urinary N-Telopeptide
Description: Samples for measurement of urinary N-telopeptide were collected at baseline prior to initiation of enzalutamide administration and at Week 41.
Time Frame: Baseline, Week 41
Population: Participants who received any amount of enzalutamide and had urinary N-telopeptide measurements at baseline and at Week 41.
Measure: Mean (Standard Deviation); unit: mmol/mmol creatinine
Arm/Group | Enzalutamide
Number analyzed (Participants) | 11
mmol/mmol creatinine | -2.00 (22.414)

13. Secondary Outcome: Change From Baseline in Urinary N-Telopeptide
Description: Samples for measurement of urinary N-telopeptide were collected at baseline prior to initiation of enzalutamide administration and at Week 49.
Time Frame: Baseline, Week 49
Population: Participants who received any amount of enzalutamide and had urinary N-telopeptide measurements at baseline and at Week 49.
Measure: Mean (Standard Deviation); unit: mmol/mmol creatinine
Arm/Group | Enzalutamide
Number analyzed (Participants) | 11
mmol/mmol creatinine | -2.36 (26.526)

14. Secondary Outcome: Change From Baseline in Urinary N-Telopeptide
Description: Samples for measurement of urinary N-telopeptide were collected at baseline prior to initiation of enzalutamide administration and at Week 57.
Time Frame: Baseline, Week 57
Population: Participants who received any amount of enzalutamide and had urinary N-telopeptide measurements at baseline and at Week 57.
Measure: Mean (Standard Deviation); unit: mmol/mmol creatinine
Arm/Group | Enzalutamide
Number analyzed (Participants) | 6
mmol/mmol creatinine | -9.33 (37.824)

15. Secondary Outcome: Change From Baseline in Urinary N-Telopeptide
Description: Samples for measurement of urinary N-telopeptide were collected at baseline prior to initiation of enzalutamide administration and at Week 65.
Time Frame: Baseline, Week 65
Population: Participants who received any amount of enzalutamide and had urinary N-telopeptide measurements at baseline and at Week 65.
Measure: Mean (Standard Deviation); unit: mmol/mmol creatinine
Arm/Group | Enzalutamide
Number analyzed (Participants) | 6
mmol/mmol creatinine | 17.67 (17.131)

ADVERSE EVENTS:
Arm/Group | Enzalutamide
Serious Adverse Events (participants affected / at risk) | 13/60
Other Adverse Events (participants affected / at risk) | 59/60
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Enzalutamide (N=60)
Angina pectoris (Cardiac disorders) | 1
Bundle branch block left (Cardiac disorders) | 1
Myocardial infarction (Cardiac disorders) | 1
Sinus bradycardia (Cardiac disorders) | 1
Small intestinal obstruction (Gastrointestinal disorders) | 1
Fatigue (General disorders) | 1
Urinary tract infection (Infections and infestations) | 2
Urosepsis (Infections and infestations) | 2
Periorbital cellulitis (Infections and infestations) | 1
Fall (Injury, poisoning and procedural complications) | 1
Incisional hernia (Injury, poisoning and procedural complications) | 1
Postoperative wound complication (Injury, poisoning and procedural complications) | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1
Embolic stroke (Nervous system disorders) | 1
Third nerve disorder (Nervous system disorders) | 1
Spinal cord compression (Nervous system disorders) | 1
Transient ischaemic attack (Nervous system disorders) | 1
Hydronephrosis (Renal and urinary disorders) | 1
Urinary retention (Renal and urinary disorders) | 1
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Enzalutamide (N=60)
Fatigue (General disorders) | 43
Anorexia (Metabolism and nutrition disorders) | 17
Constipation (Gastrointestinal disorders) | 17
Arthralgia (Musculoskeletal and connective tissue disorders) | 16
Back pain (Musculoskeletal and connective tissue disorders) | 14
Oedema peripheral (General disorders) | 14
Nausea (Gastrointestinal disorders) | 11
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 10
Hot Flush (Vascular disorders) | 9
Bone pain (Musculoskeletal and connective tissue disorders) | 8
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 8
Dysgeusia (Nervous system disorders) | 7
Insomnia (Psychiatric disorders) | 7
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 7
Pollakiuria (Renal and urinary disorders) | 6
Urinary incontinence (Renal and urinary disorders) | 6
Blood alkaline phosphatase increased (Investigations) | 5
Cough (Respiratory, thoracic and mediastinal disorders) | 5
Pain in extremity (Musculoskeletal and connective tissue disorders) | 5
Depression (Psychiatric disorders) | 4
Dry skin (Skin and subcutaneous tissue disorders) | 4
Headache (Nervous system disorders) | 4
Muscle spasms (Musculoskeletal and connective tissue disorders) | 4
Vomiting (Gastrointestinal disorders) | 4
Abdominal pain (Gastrointestinal disorders) | 3
Contusion (Injury, poisoning and procedural complications) | 3
Dyspepsia (Gastrointestinal disorders) | 3
Fall (Injury, poisoning and procedural complications) | 3
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 3
Pain (General disorders) | 3
Peripheral sensory neuropathy (Nervous system disorders) | 3
Rash (Skin and subcutaneous tissue disorders) | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
PI agrees not to independently publish the results before the publication of the multi-center PI paper. Sponsor shall review and comment 30 days prior to submission or disclosure. If publication or disclosure contains Sponsor Confidential Information, other than Study Data, PI agrees to remove Confidential Information from publication or disclosure. Sponsor may request that PI delay such publication for an additional 60 days to protect the patentability of any Invention described.